CLINICAL TRIAL: NCT04405362
Title: Consequences of the QUARANTINE Relating to the COvid-19 Epidemic on the Mental Health of the Patients Followed in PSYchiatry
Acronym: QUARCOPSY
Status: Withdrawn | Type: Observational
Why Stopped: NO INCLUSION
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_39; 2020-A01186-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV 2; Traumatic Stress Disorder
Keywords: COVID-19; quarantine; Psychiatric Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quarantine related to the Covid-19 pandemic has begun on the 03/17/2020 in France. Quarantine has already be linked to pejorative effects on mental health. In this study, we aim to evaluated PTSD symptoms of patients already followed by a psychiatrist during quarantine, one month and 3 months after inclusion. It will be also evaluate various psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients already followed in psychiatry before quarantine by one of the psychiatrists subscribed to L'Encéphale online.

Exclusion Criteria:

* Refusal to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with psychotic disorder, mood disorders, labile emotional personality disorder, anxiety disorders and somatoform disorders
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with post-traumatic stress disorder (PTSD) defined by a total score on PCL-5 ≥ 31 at the time of quarantine | at inclusion
  PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-5). The PCL-5 is an instrument that consists of 20 items rated from 0 to 4 to obtain a score from 0 to 80. A score greater than or equal to 31-33 defines the presence of posttraumatic stress disorder.
Number of patients with post-traumatic stress disorder (PTSD) defined by a total score on PCL-5 ≥ 31 at the time of quarantine | at 1 month after inclusion
  PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-5). The PCL-5 is an instrument that consists of 20 items rated from 0 to 4 to obtain a score from 0 to 80. A score greater than or equal to 31-33 defines the presence of posttraumatic stress disorder.
Number of patients with post-traumatic stress disorder (PTSD) defined by a total score on PCL-5 ≥ 31 at the time of quarantine | at 3 months after inclusion
  PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-5) (6). The PCL-5 is an instrument that consists of 20 items rated from 0 to 4 to obtain a score from 0 to 80. A score greater than or equal to 31-33 defines the presence of posttraumatic stress disorder.

SECONDARY OUTCOMES:
IES-R (Impact of Events Scale Revised) | at inclusion, then at 1 month and 3 months after inclusion
  This self-questionnaire is intended to measure subjective post-traumatic stress after a traumatic situation (within 7 days) but is not a diagnostic tool. It includes 22 items rated from 0 (not at all) to 4 (extremely). There are 3 sub-scales:
  * an avoidance subscale (items 5, 7, 8, 11, 12, 13, 17, 22): the sum of the scores on each of these items ranges from 0 to 35;
  * Memory intrusion subscale (items 1, 2, 3, 6, 9, 14, 16 and 20): the sum of the scores on each of these items ranges from 0 to 40;
  * a Hyperarousal/High Neurovegetative Activation subscale (items 4, 10, 15, 18, 19 and 21): the sum of the scores on each of these items ranges from 0 to 35.
  A total score of at least 22 suggests the presence of significant symptoms of acute stress. A score of 36 and above suggests the presence of post-traumatic stress disorder.
Presence of suicidal ideation during the past month at the different times of the study | at inclusion, then at 1 month and 3 months after inclusion
  closed-ended question: Yes /No
Total score at GHQ-28 (General Health Questionnaire) | at inclusion, then at 1 month and 3 months after inclusion
  questionnaire with a 28 item scaled and assesses somatic symptoms, anxiety and insomnia, social dysfunction and severe depression that ranges from a 'better/healthier than normal' option, through a 'same as usual' and a 'worse/more than usual' to a 'much worse/more than usual' option. The exact wording will depend upon the particular nature of the item.
Total score at BDI (Beck Depression Inventory) | at inclusion, then at 1 month and 3 months after inclusion
  13 questions rated from 0 to 3 to obtain a score from 0 to 39 The higher the score, the greater the symptomatology: 0 to 3 (no depression), 4 to 7 (mild depression), 8 to 15 (depression of moderate to moderate intensity), greater than 16 (severe depression).
Total score at ISI (Insomnia Severity Index) | at inclusion, then at 1 month and 3 months after inclusion
  7 questions rated from 0 to 4 to obtain a score from 0 to 28 The higher the score, the greater the symptomatology: 0 to 7 (no insomnia), 8 to 14 (mild insomnia), 15 to 21 (moderate insomnia), 22 to 28 (severe insomnia).
Changes in alcohol and/or cannabis consumption during and at the end of the quarantine period | at inclusion, then at 1 month and 3 months after inclusion
Total score Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | at inclusion, then at 1 month and 3 months after inclusion
  It's a Likert scale from 14 to 70. The higher the score, the higher the level of well-being.
Socio-demographic factors significantly associated with all scores | at inclusion, then at 1 month and 3 months after inclusion
  Socio-demographic factors, linked to medical history and the experience of the epidemic.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Leroy, MD, Principal Investigator — University Hospital, Lille